CLINICAL TRIAL: NCT02574897
Title: Evaluating the Ability of Electronic Patient Symptom Reporting to Reduce Symptom Burden During Hospitalization for Intensive Chemotherapy
Brief Title: The Ability of Electronic Patient Symptom Reporting to Reduce Symptom Burden During Hospitalization for Chemotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: LCCC 1404
Record Dates: First submitted 2015-02-20; First posted 2015-10-14 (Estimated); Last update posted 2018-03-22 (Actual); Status verified 2018-03

CONDITIONS: Stem Cell Transplantation, Hematopoietic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Electronic Symptom Survey (Experimental): Patients randomized to the intervention arm will fill out the daily PRO-CTCAE electronic symptom survey. The intervention consists of sending the results of the surveys in the intervention arm to the clinical care team. The four symptom-specific PROMIS subsets (Anxiety, Depression, Fatigue, and Sleep Disturbance) will be filled out weekly while patients are admitted to the hospital. Patients will again complete the 6 minute walk distance testing, HRQoL surveys, and PASS assessment at the time of discharge. Patients in the intervention arm will complete a satisfaction survey at discharge. HRQoL (by mail) and PASS (by telephone) will be assessed for a third time 30 days after discharge.
  Interventions: Other: Electronic symptom survey
- Blinded Electronic Symptom Survey (Active Comparator): Patients in the control arm will only fill out the symptom survey at the time of admission and days 7, 10, and 14. The results of symptom surveys from the patients in the control arm will not be sent to providers, but will be used for data analysis purposes only. The four symptom-specific PROMIS subsets (Anxiety, Depression, Fatigue, and Sleep Disturbance) will be filled out weekly while patients are admitted to the hospital. Patients will again complete the 6 minute walk distance testing, HRQoL surveys, and PASS assessment at the time of discharge. HRQoL (by mail) and PASS (by telephone) will be assessed for a third time 30 days after discharge.
  Interventions: Other: Blinded Electronic Symptom Survey

INTERVENTIONS:
Other: Electronic symptom survey — Standard of care plus daily electronic symptom surveys, the results of which are sent to clinicians electronically.
  Other Names: Online Daily Symptom Survey
  Arms: Electronic Symptom Survey
Other: Blinded Electronic Symptom Survey — Standard of care daily clinician interviews with blinded symptom surveys
  Arms: Blinded Electronic Symptom Survey

SUMMARY:
The purpose of this randomized trial will evaluate whether providing clinicians with daily reports from a well-validated, standardized, patient-centered electronic symptom survey tool (PRO-CTCAE) improves symptom burden in patients undergoing high-dose chemotherapy. Adult inpatients at UNC undergoing high-dose chemotherapy for preparative chemotherapy prior to stem cell infusion. Participants will be randomized into one of two arms: (1) a control arm with standard of care daily clinician interviews or (2) standard of care plus daily electronic symptom surveys, the results of which will be sent to clinicians electronically.

DETAILED DESCRIPTION:
The primary objective of the study is to compare peak symptom burden between the two study arms (autologous transplant vs. allogeneic transplant). Peak symptom burden will also be compared between the two study arms within both subgroups of patients (myeloablative vs. reduced intensity conditioning). Secondary outcomes that will also be compared between the two arms include: changes in patient-reported quality of life, time to supportive care treatment changes, length of hospital stay, thirty day readmission rate after discharge, days alive and out of the hospital in the 100 days since admission, and overall survival. Additionally, measures of physical activity will be captured through physiological monitoring in order to explore associations with patient-reported symptom measures. Patient and clinician satisfaction will also be evaluated.

In this study, the investigators will use an electronic survey to assess 16 patient-reported symptoms to calculate a symptom score that may range from 0-61 each day. This symptom score represents the symptom burden for the patient on that particular day. Symptom burden is anticipated to peak between days 7 and 14, so the investigators will define peak symptom burden as the average of the symptom scores on days 7, 10 and 14. In both arms, symptoms will be assessed on these days in order to compare peak burden.

ELIGIBILITY:
Inclusion Criteria:

* Verification of access to a functioning email account
* >= 18 years of age
* <= 75 years of age
* Able to read in English
* Assessed as competent based on discretion of study personnel
* Willing and able to provide signed, informed consent

Exclusion Criteria:

* Concurrent participation in LCCC1234

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2014-07; Primary Completion 2017-06-30 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Average peak symptom burden in the intervention group versus the control group | Measured by comparing the average PRO-CTCAE scores from Day+7, Day+10, and Day+14 in the intervention compared to the control group
  Peak symptom burden is defined as the average symptom score on chemotherapy days+7, +10, and +14 (relative to transplant day 0) as measured by the PRO-CTCAE. There are 16 items on the PRO-CTCAE questionnaire. Fifteen items are worth 0-4 points each and one item is worth 0-1 point. This translates to a symptom score range of 0-61 per day, which will be averaged over the three days. The outcome is the comparison of average peak symptom burden scores between the two groups.

CONTACTS AND LOCATIONS:
Overall Officials: Ashley L Bryant, PHD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (1):
- Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bryant AL, Coffman E, Phillips B, Tan X, Bullard E, Hirschey R, Bradley J, Bennett AV, Stover AM, Song L, Shea TC, Wood WA. Pilot randomized trial of an electronic symptom monitoring and reporting intervention for hospitalized adults undergoing hematopoietic stem cell transplantation. Support Care Cancer. 2020 Mar;28(3):1223-1231. doi: 10.1007/s00520-019-04932-9. Epub 2019 Jun 20. PMID 31222392